CLINICAL TRIAL: NCT00460083
Title: A Randomized, Double-Blinded Study of Epiceram Versus Elidel in Pediatric Subjects With Mild to Moderate Atopic Dermatitis
Brief Title: Epiceram Versus Elidel for Treatment of Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ceragenix Pharmaceuticals (Industry)
Responsible Party: Sr. Vice President, Research & Development, Ceragenix Pharmaceuticals Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CGXP - 060674/ IRB00002569
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Last update posted 2008-02-06 (Estimated); Status verified 2008-02

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; eczema; dermatitis; skin barrier; barrier repair; ceramide; physiologic lipid; pruritus; Elidel; Epiceram; topical steroid
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Dermatitis; Pruritus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elidel(r) (Active Comparator)
  Interventions: Drug: Elidel(R) (pimecrolimus 1%)
- Epiceram(r) (Experimental)
  Interventions: Device: EpiCeram(R) -ceramide based barrier repair cream

INTERVENTIONS:
Drug: Elidel(R) (pimecrolimus 1%)
  Arms: Elidel(r)
Device: EpiCeram(R) -ceramide based barrier repair cream
  Arms: Epiceram(r)

SUMMARY:
Atopic dermatitis (AD) is a common skin disease that has increased in prevalence worldwide two- to threefold over the last 50 years. Epiceram, a newly FDA-approved medical device is a topical barrier repair cream designed to deliver special epidermal lipids to the top layers of the skin in order to correct skin barrier abnormalities found in atopic dermatitis. Epiceram does not contain corticosteroids or other conventional anti-inflammatory components and represents a novel class of skin barrier repair therapy for inflammatory skin disease.

The objective of this study is to determine whether Epiceram is a safe and effective therapy for mild to moderate atopic dermatitis and whether it may serve as an alternative to Elidel therapy.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a common skin disease that has increased in prevalence worldwide two- to threefold over the last 50 years. Current standard of care for atopic dermatitis includes topical corticosteroids and calcineurin inhibitors, such as Elidel and Protopic. The chronic use of topical corticosteroids is limited by side effects including skin atrophy, striae, and even HPA axis suppression. The long-term effects of skin immunosuppression with calcineurin inhibitors are unknown and although not proven, a theoretical risk of skin cancer exists. Novel therapies for atopic dermatitis that avoid immunosupression are greatly needed.

Epiceram, a newly FDA-approved medical device is a topical barrier repair cream designed to deliver special epidermal lipids to the top layers of the skin in order to correct skin barrier abnormalities found in atopic dermatitis. Epiceram does not contain corticosteroids or other conventional anti-inflammatory components and represents a novel class of skin barrier repair therapy for inflammatory skin disease. The objective of this study is to determine whether Epiceram is a safe and effective therapy for mild to moderate atopic dermatitis and whether it may serve as an alternative to Elidel therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females of any race 2 - 12 years of age.
2. Diagnosis of atopic dermatitis on the basis of the criteria defined by Hanifin and Rajka (Hanifin, 1980).
3. Rajka-Langeland Severity Index score of mild to moderate (Rajka, 1989).
4. At least one antecubital or popliteal fossa must be affected at the time of enrollment to serve as a target site.

Exclusion Criteria:

1. Subjects with severe AD as determined by the Rajka-Langeland Severity Index (Rajka 1989).
2. Disease severity requiring medium-potency topical steroid medication to treat their atopic dermatitis more than 1 week per month.
3. Subjects with unstable or uncontrolled medical conditions that could require intensive treatment during the course of the study.
4. Subjects who require greater than 2.0 mg/day inhaled or intranasal corticosteroids.
5. Subjects who are currently participating in or, within the past 28 days, have participated in another study using an investigational drug.
6. Subjects with a history of allergy or hypersensitivity to Epiceram, Elidel, or ingredients therein, including fragrances.
7. Active infection of any type at the start of the study.
8. Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated.
9. Subjects must have not used any topical or systemic therapy during the washout periods.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2007-04; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
The primary efficacy outcome is the change in mean Eczema Area and Severity Index (EASI) score in both groups. | 4 weeks

SECONDARY OUTCOMES:
Percent of subjects reaching clear or almost clear on Investigator's Global Assessment (IGA) at week 4. | 4 weeks
Change in mean capacitance in lesional and nonlesional skin at target site | 4 weeks
Change in mean transepidermal water loss (TEWL) in lesional and nonlesional skin at target site | 4 weeks
Change in pruritus score measured with a visual analog scale | 4 weeks
Comparison of baseline and Week 4 Children's Dermatitis Life Quality Index (CDLQI) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eric Simpson, MD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - UCSD, San Diego, California
  - OHSU, Portland, Oregon